CLINICAL TRIAL: NCT04030065
Title: Randomized Controlled Trial to Study the Effect of Intravenous Supplementation of Omega-3 Fatty Acids on Outcome of Recipients in Living Donor Liver Transplantation (LDLT)
Brief Title: Study to Assess the Effect of Intravenous Supplementation of Omega-3 Fatty Acids on Outcome of Recipients in Living Donor Liver Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Vivek Rajendran, Senior Resident, Department of HPB surgery and Liver transplantation, Institute of Liver and Biliary Sciences, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ILBS-livertransplant-01
Record Dates: First submitted 2019-07-11; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm - omega 3 fatty acid (Experimental)
  Interventions: Drug: Omega 3 fatty acid
- Control Arm - No intervention (No Intervention)

INTERVENTIONS:
Drug: Omega 3 fatty acid — 10% Omega-3 fatty acid oil will be supplemented in intravenous form from preoperative day 1, intra-operatively (anytime during surgery before reperfusion of graft) and from post operative day 1 to day 5 in the study group. The preparation used will be 100 ml injection which contains 10 gm of Omega 3 fatty acids.
  Arms: Experimental Arm - omega 3 fatty acid

SUMMARY:
In this study, the investigators aim to analyse the effect of Omega 3 fatty acid supplementation on recipients undergoing living donor liver transplantation. In Group A, the patients receive Omega 3 fatty acid on preoperative day 1, intraoperatively and up to day 5 post operatively; and the effect of omega 3 fatty acid supplementation on early allograft dysfunction, its correlation with occurrence of postoperative complications and liver regeneration measured by CT volumetry on Day 7. Group B, the patients are controls for the study and hence attempt to find out the effect of omega 3 fatty acid supplementation on outcome of recipients of Living donor liver transplantation. the investigators will analyse the data and elucidate the value of omega 3 fatty acid supplementation in reducing the occurrence of early allograft dysfunction , complications and effect on liver regeneration in recipients of Living donor liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All elective liver transplant recipients
* Adult patients
* Those who consent

Exclusion Criteria:

* Liver transplantation for fulminant hepatic failure
* Re-transplantation
* Known allergy to the study emulsion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2018-12-02 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Early Allograft Dysfunction | Post operative day 7
  To study the correlation with early allograft dysfunction using definition of early allograft dysfunction based on laboratory parameters (presence of one or more of the following : bilirubin >or=10mg/dL on day 7, international normalized ratio >or=1.6 on day 7, and alanine or aspartate aminotransferases >2000 IU/L within the first 7 days)

SECONDARY OUTCOMES:
Liver function test - trend | Till period of hospital stay, average of 1 month
  To study the correlation between supplementation of omega-3 fatty acids and trend in post-operative LFTs
Complications | Till period of hospital stay, average of 1 month
  Post-operative complications
ICU and hospital stay | Till period of hospital stay, average of 1 month
  To determine the total hospital stay and ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Viniyendra Pamecha, Professor, Study Chair — Professor and head , Department of HPB surgery and liver Transplantation, ILBS, New Delhi
Locations (1):
- Institute of liver and biliary Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided